CLINICAL TRIAL: NCT02395497
Title: Human Penile Allotransplantation
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00089306
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2025-07-07 (Actual); Status verified 2025-07

CONDITIONS: Amputation; Wounds and Injuries; Amputation, Traumatic; Urologic Surgical Procedures, Male; Amputation, Traumatic/Surgery; Penis/Transplantation; Penis/Surgery; Penis/Injuries; Congenital Anomaly, Male Genitalia
Keywords: Penile Transplant; Vascularized Composite Allotransplantation (VCA); Composite Tissue Allotransplantation (CTA); Penis; Amputation; Immunosuppression; Composite Tissue; Male; Humans; Allotransplantation; Micropenis; Severely Aambiguous Male Genitalia; congenital/birth defect
MeSH Terms: conditions — Wounds and Injuries; Amputation, Traumatic; Congenital Abnormalities; Penis agenesis | interventions — Antibodies, Monoclonal; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: Transplantation (Experimental): Penile transplantation with an immunomodulatory protocol consisting of monoclonal antibody induction therapy of humanized anti CD52 followed by donor bone marrow infusion and tacrolimus monotherapy.
  Interventions: Biological: Monoclonal Antibody (Humanized Anti-CD52); Drug: Tacrolimus; Procedure: Penile Allotransplantation

INTERVENTIONS:
Biological: Monoclonal Antibody (Humanized Anti-CD52)
Drug: Tacrolimus
Procedure: Penile Allotransplantation

SUMMARY:
Injuries to the genitalia are of concern to the military with emphasis placed on the surgical reconstruction and psychological health of these Wounded Warriors. However, despite significant surgical advances in microvascular surgery and autologous free tissue transfer, conventional reconstructions cannot truly replace the complicated structures and functions of the penis including the urethra, erogenous sensation, and erectile corporal bodies. Conventional reconstruction poses several challenges: patients may not have sufficient donor tissue due to other injuries or previous surgery; multiple operations are often needed to restore the neophallus; the final reconstruction only approximates the penis' native form; recreating the urethra is challenging and the new urethra is prone to stricture and fistula formation; the erectile function necessary for sexual intercourse is often lacking; and insufficient protective sensation can lead to penile implant extrusion, infection, subsequent explantation or loss of the reconstruction.

The investigators propose this clinical trial to determine functional outcomes and quality of life for Wounded Warriors and civilians who choose to undergo penile allotransplantation. The investigators will combine extensive experience performing total penile reconstruction in a large population affected by congenital, traumatic, and therapeutically extirpated Genitourinary deformities and expertise in reconstructive transplantation using an immunomodulatory protocol to for this study. The investigators anticipate penile transplantation can potentially replace "like with like," restoring the appearance, anatomy, and function of the recipient in a manner far superior to autologous reconstruction. This project will establish the ability to perform penile allotransplantation using an immunomodulatory protocol and will compare outcomes with conventional phalloplasty patient results.

Study Design: This is a non-randomized subject self-controlled clinical trial to implement a cell-based immunomodulatory protocol for penile allotransplantation. An intermediate deliverable is achieving allograft survival and functional return with reduced dosing/frequency of maintenance immunosuppression on steroid-free monotherapy (tacrolimus) immunosuppression. The long-term deliverable and goal is to demonstrate superior outcomes when compared to satisfaction and QOL in conventional phalloplasty patients 12-60 months post-transplant.

DETAILED DESCRIPTION:
Specific Aims: 1) To assess the feasibility and function of penile allotransplantation in Wounded Warriors and civilians who have lost their penis due to battle or traumatic injury, using an immunomodulatory protocol to reduce immunosuppression; 2) To assess pre-to-post changes in QOL in patients who undergo penile allotransplantation.

ELIGIBILITY:
Donor Inclusion Criteria:

* Males aged 16 - 65 years.
* Brain dead meeting the criteria for Determination of Death.
* Family consent for penile graft donation.
* Stable donor (i.e., does not require excessive vasopressors to maintain blood pressure).
* Same blood type as recipient.
* Negative lymphocytotoxic crossmatch.
* Accurately matched for skin tone

Recipient Inclusion Criteria:

* Males of any race, color or ethnicity; aged 18-69 years.
* Recent (≥6 months) or remote (i.e., several decades) penile injury resulting in the loss of ≥75% of the phallus.
* Penectomy secondary to penile cancer
* Penile Cancer Survivors > 5 years
* Micropenis associated with congenital/birth defect and severely ambiguous male genitalia
* Must have completed a clinic appointment with one of the study surgeons to discuss all penile reconstructive options.
* Completes the protocol informed consent form(s).
* No co-existing medical condition which, in the opinion of the study team, could affect the immunomodulatory protocol, surgical procedure, or functional results (If the condition is amenable to treatment, the study team must agree that said condition should not significantly enhance the surgical risks of penile transplantation.).
* No co-existing psycho-social problems (i.e., alcoholism, drug abuse).
* Negative for malignancy for past 5 years.
* Negative for HIV at transplant.
* Negative crossmatch with donor.
* Consents to sample (i.e., skin biopsy) collection and storage and bone marrow infusion as part of the treatment regimen.
* USA citizen or equivalent.
* Patient agrees to comply with the protocol and states a dedication to the immunomodulatory treatment regimen.

Recipient and Donor Exclusion Criteria:

* Untreated sepsis.
* HIV (active or seropositive).
* Active tuberculosis.
* Active Hepatitis B infection.
* Hepatitis C.
* Viral encephalitis.
* Toxoplasmosis.
* Malignancy (within past 5 years).
* Current/recent (within 3 months of donation/screening consent) IV drug abuse.
* Paralysis of ischemic or traumatic origin.
* Inherited peripheral neuropathy.
* Infectious, post infectious, or inflammatory (axonal or demyelinating) neuropathy.
* Toxic neuropathy (i.e. heavy metal poisoning, drug toxicity, industrial agent exposure).
* Mixed connective tissue disease.
* Severe deforming rheumatoid or osteoarthritis in the limb.

Donor Only Exclusion Criteria:

* Evidence of active herpes simplex virus-2 (HSV-2) infection.
* Tattoos: non-professional tattoo within the last 6 months, or personally identifiable tattoo (i.e., donor name) on potential transplant.

Recipient Only Exclusion Criteria:

* Conditions that, in the opinion of the study team, may impact the immunomodulatory protocol potentially exposing the recipient to an unacceptable risk under immunosuppressive treatment.
* Sensitized recipients with high levels (50%) of panel-reactive human leukocyte antigen (HLA) antibodies.
* Conditions that may impact the success of the surgical procedure or increase the risk of postoperative complications including inherited coagulopathies like Hemophilia, Von-Willebrand's disease, Protein C and S deficiency, Thrombocythemias, Thalassemias, Sickle Cell disease, etc.
* Conditions that may impact functional outcomes including Lipopolysaccharidosis and amyloidosis (may impact nerve regeneration).
* Patients considered psychologically/psychiatrically unsuitable.

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2034-06 (Estimated); Study Completion 2039-06 (Estimated)

PRIMARY OUTCOMES:
Allograft Survival | Transplantation through end of study period (up to 5 years)
  use an immunomodulatory protocol to reduce immunosuppression. Post-operative allograft survival will be assessed by various clinical measures including: physical assessments, imaging assessments (ultrasound, CT angiography, magnetic resonance (MR) Neurography and MRI) immune monitoring (screen patient sera for donor specific antibodies), hematologic and metabolic tests, viral tests, chimerism tests, and skin biopsies

SECONDARY OUTCOMES:
Quality of Life (QOL) as assessed by Brief Symptom Inventory | Transplantation through end of study period ( 5 years)
  Brief Symptom Inventory questionnaire evaluates psychological distress and psychiatric disorders. It consists of 53-item self-report inventory in which participants rate the extent to which they have been bothered. 5-point rating scale, 0 indicating not at all bothered to 4 extremely bothered.
QOL as assessed by Affect Balance Scale (ABS) | Transplantation through end of study period (up to 5 years)
  ABS is a 10-item questionnaire that assess positive and negative affect as indicators of life satisfaction and/or well-being. Score range from 0-4. 0 indicating the feeling never affected to 4, where the feeling is affected always.
QOL as assessed by NEO Five-Factor Inventory Scale (NEO-FFI) | Transplantation through end of study period (up to 5 years)
  NEO-FFI is used to examine personality traits. Questions consists of 60 items. Items are scored from Strongly disagree to Strongly agreed
QOL as assessed by the International Index of Erectile Function (IIEF) | Transplantation through end of study period (up to 5 years)
  A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
Psychosexual Measures assessed by Self-Esteem and Relationship (SEAR) questionnaire | Transplantation through end of study period ( 5 years)
  14 item questionnaire where responses are scored from 1-5. Response of 1 indicating almost never/never to 5 indicating almost always/always
T0 asses Erection Hardness Score (EHS) | Transplantation through end of study period ( 5 years)
  EHS rates the hardness of erection on a scale of one to four, with four being the maximal score.
Modified Sexual Life Quality Questionnaire-Quality of Life (mSLQQ- QoL) | Transplantation through end of study period ( 5 years)
  Used to validate as a tool for evaluating sexual QoL. mSLQQ is measured from score of 0 to 8. 0 indicates a low score compare to 8, indicating high. A score of 4 indicates, nothing has been changed.
Psychological Measures by Satisfaction with Life Scale (SWLS) | Transplantation through end of study period ( 5 years)
  SWLS is a measure of life satisfaction. Uses scale to rate from 1-7, Where 1 indicates Strongly disagree to 7 indicating strongly agree.
Brief Pain Inventory (Short Form) ) (BPISF) | Transplantation through end of study period ( 5 years)
  BPISF assesses the severity of pain and its impact on functioning. It is scored from 0 to 10, 0 indicating no pain, does not interfere to 10 indicating pain as bad as you can imagine, completely interferes.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Redett, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Schneeberger S, Gorantla VS, Brandacher G, Zeevi A, Demetris AJ, Lunz JG, Metes DM, Donnenberg AD, Shores JT, Dimartini AF, Kiss JE, Imbriglia JE, Azari K, Goitz RJ, Manders EK, Nguyen VT, Cooney DS, Wachtman GS, Keith JD, Fletcher DR, Macedo C, Planinsic R, Losee JE, Shapiro R, Starzl TE, Lee WP. Upper-extremity transplantation using a cell-based protocol to minimize immunosuppression. Ann Surg. 2013 Feb;257(2):345-51. doi: 10.1097/SLA.0b013e31826d90bb. PMID 23001085
- [Background] Bluebond-Langner R, Redett RJ. Phalloplasty in complete aphallia and ambiguous genitalia. Semin Plast Surg. 2011 Aug;25(3):196-205. doi: 10.1055/s-0031-1281489. PMID 22851911
- [Background] Massanyi EZ, Gupta A, Goel S, Gearhart JP, Burnett AL, Bivalacqua TJ, Redett RJ. Radial forearm free flap phalloplasty for penile inadequacy in patients with exstrophy. J Urol. 2013 Oct;190(4 Suppl):1577-82. doi: 10.1016/j.juro.2012.12.050. Epub 2012 Dec 25. PMID 23270911
- [Background] Tuffaha SH, Sacks JM, Shores JT, Brandacher G, Lee WPA, Cooney DS, Redett RJ. Using the dorsal, cavernosal, and external pudendal arteries for penile transplantation: technical considerations and perfusion territories. Plast Reconstr Surg. 2014 Jul;134(1):111e-119e. doi: 10.1097/PRS.0000000000000277. PMID 24622570
- [Background] Schneeberger S, Landin L, Jableki J, Butler P, Hoehnke C, Brandacher G, Morelon E; ESOT CTA Working Group. Achievements and challenges in composite tissue allotransplantation. Transpl Int. 2011 Aug;24(8):760-9. doi: 10.1111/j.1432-2277.2011.01261.x. Epub 2011 May 9. PMID 21554424